CLINICAL TRIAL: NCT06386328
Title: An Open-label, Randomized, Single-dose, 2-sequence, 2-period, Crossover, Phase 1 Study to Evaluate the Food Effect on the Pharmacokinetics and Safety of CKD-378 in Healthy Volunteers
Brief Title: A Clinical Trial to Evaluate the Food Effect of CKD-378
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A129_03FDI2317
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-05

CONDITIONS: Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): * Period 1: A single oral dose of 2 tablets(CKD-378) under fasting condition
  * Period 2: A single oral dose of 2 tablets(CKD-378) under fed condition
  Interventions: Drug: CKD-378, QD, PO
- Sequence 2 (Experimental): * Period 1: A single oral dose of 2 tablets(CKD-378) under fed condition
  * Period 2: A single oral dose of 2 tablets(CKD-378) under fasting condition
  Interventions: Drug: CKD-378, QD, PO

INTERVENTIONS:
Drug: CKD-378, QD, PO — CKD-378, QD, PO

SUMMARY:
A clinical trial to evaluate the food effect of CKD-378

DETAILED DESCRIPTION:
An open-label, randomized, single-dose, 2-sequence, 2-period, crossover, phase 1 study to evaluate the food effect on the pharmacokinetics and safety of CKD-378 in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult aged ≥ 19 at screening
2. Body mass index (BMI) of 18.0 kg/m2 or more and less than 30.0kg/m2 and Body weight ≥ 50kg
3. Those who do not have congenital or chronic diseases and have no pathological symptoms or findings as a result of medical examination
4. A person who is deemed suitable as a subject as a result of screening such as clinical laboratory examination (hematology, blood chemistry, serological tests, urinalysis, etc.), electrocardiogram examination, etc.
5. A person who has received a sufficient explanation of the purpose and contents of the clinical trial and has agreed in writing voluntarily to participate in the clinical trial
6. A person who has agreed to use appropriate contraception and not donate sperm or eggs until 1 week after the first administration of the drug and the last administration of the drug

Exclusion Criteria:

1. Those who have taken a drug known to significantly induce or inhibit drug metabolizing enzymes within 30 days before the first administration of investigational product, or who have taken drug that may interfere with this investigational product within 10 days
2. Those with a history of regular alcohol intake before the first administration of investigational product

   * More than 21 drinks/week for men
   * More than 14 drinks/week for women
3. Those who have taken other investigational product within 6 months before the first administration of the investigational product
4. Those who have donated whole blood within 8 weeks or donated component blood within 2 weeks or received blood transfusion within 4 weeks before the first administration of the investigational product
5. Those with a history of gastrointestinal diseases or surgery (except simple appendicectomy, hernia surgery) that may affect drug absorption ruler
6. Those who have following diseases

   * Patients with hypersensitivity to the ingredient of an investigational drug or to biguanide drugs
   * Patients with moderate and severe renal impairment, end-stage renal disease or dialysis
   * Patients with acute conditions that may affect renal function
   * Patients with acute or chronic metabolic acidosis and patients with a history of ketoacidosis
   * Diabetic precoma patient
   * Patients with acute and unstable heart failure
   * Patients receiving tests using intravenous radioactive iodine contrast material
   * Patients with severe infections or severe traumatic systemic disorders
   * Patients scheduled for surgery
   * Patients with malnutrition, starvation, weakness, pituitary dysfunction, or adrenal dysfunction
   * Patients with gastrointestinal disorders
7. A history of clinically significant psychiatric disease
8. Those who are judged by the investigator for reason other than the above selection/exclusion criteria and are judged unsuitable for participation in the study
9. Woman who are suspected of being pregnant or breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-378 | Pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 24, 32, 48 hours
  Area under the concentration-time curve time zero to time
Cmax of CKD-378 | Pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 24, 32, 48 hours
  Maximum plasma concentration of the drug

CONTACTS AND LOCATIONS:
Locations (1):
- Gimpo Woori hospital, Gimpo-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No